CLINICAL TRIAL: NCT07231822
Title: The Investigation of the Effectiveness of Virtual Reality Applications in Postmenopausal Osteoporosis Patients: A Randomized Controlled Trial
Brief Title: The Investigation of the Effectiveness of Virtual Reality Applications in Postmenopausal Osteoporosis Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kirsehir Ahi Evran Universitesi (Other)
Responsible Party: Principal Investigator, İrem CANLI, Research Assistant, Kirsehir Ahi Evran Universitesi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 23591230588?
Record Dates: First submitted 2025-11-14; First posted 2025-11-17 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-11

CONDITIONS: Osteoperosis
Keywords: Postmenopausal osteoporosis; Virtual reality; balance
MeSH Terms: conditions — Osteoporosis, Postmenopausal

STUDY DESIGN:
Intervention Model Description: Randomized dontrolled trial
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Experimental): Traditional treatment will consist of posture exercises aimed at ensuring proper posture, strengthening exercises, balance exercises, patient education aimed at preventing falls and fractures, aerobic exercises, and interventions aimed at controlling acute and chronic pain and restoring independence in daily living activities.
  Interventions: Other: Conventional treatment
- Virtual Reality Group (Experimental): Virtual reality applications will consist of videos and video-based games (exergames). Should an application pose a risk to patients, the programme will be reviewed.
  Interventions: Other: Conventional treatment; Other: Virtual reality treatment

INTERVENTIONS:
Other: Conventional treatment — Traditional treatment will consist of posture exercises aimed at ensuring proper posture, strengthening exercises, balance exercises, patient education aimed at preventing falls and fractures, aerobic exercises, and interventions aimed at controlling acute and chronic pain and restoring independence in daily living activities.
Other: Virtual reality treatment — Virtual reality applications will consist of videos and video-based games (exergames). Should an application pose a risk to patients, the programme will be reviewed.
  Arms: Virtual Reality Group

SUMMARY:
Osteoporosis is a progressive disease characterised by a decrease in bone mass, deterioration in bone microarchitecture, and increased fragility. Etiologically, it is divided into two types: primary (postmenopausal and senile) and secondary. Postmenopausal women are particularly at high risk; it is seen in more than 80% of women over the age of 50 and in almost all individuals over the age of 75. With menopause, bone mineral density decreases, which negatively affects neuromuscular functions, leading to balance disorders, decreased walking speed, and an increased risk of falls. Falls are the primary cause of osteoporotic fractures and result in functional loss, morbidity, mortality, and increased healthcare costs. Exercise is effective in reducing bone loss; in recent years, therapeutic virtual reality and exercise games (exergames) have come to the fore. However, the literature on the effectiveness of these applications in postmenopausal osteoporosis patients is limited. The aim of this study is to investigate the effects of virtual reality applications on balance, quality of life, and fall risk and to compare them with a control group.

DETAILED DESCRIPTION:
According to the World Health Organisation's definition, osteoporosis is characterised as a progressive disease involving a decrease in bone mass, deterioration in bone microarchitecture, and an increase in bone fragility. Osteoporosis is classified into two types based on aetiological factors: primary and secondary. Primary osteoporosis is subdivided into postmenopausal and senile osteoporosis, while the aetiology of secondary osteoporosis is unclear. Although osteoporosis can affect people of all ages, postmenopausal women are a particularly high-risk group for developing osteoporosis. Osteoporosis is seen in more than 80% of women over the age of 50 and in almost all women and men over the age of 75. Postmenopausal osteoporosis is the most common form of the disease. With the onset of menopause, a progressive decrease in bone mineral density is observed. This decrease in bone mineral density negatively affects the neuromuscular system. Neuromuscular dysfunction in patients with postmenopausal osteoporosis leads to a decrease in the ability to stand, impaired dynamic balance, and an increased risk of falling due to a decrease in walking speed. Falls are a significant risk factor in the development of osteoporotic fractures. The occurrence of osteoporosis-related fractures can lead to a decrease in functional capacity, an increase in morbidity and mortality rates, and higher healthcare costs. Exercise has a positive effect on reducing bone mineral density loss. However, advances in technology have also increased the availability of video games for therapeutic purposes. Virtual reality or exergame applications that incorporate video games have become a new trend in response to the global challenges of ageing. However, there is limited literature investigating the effectiveness of virtual reality applications in postmenopausal osteoporosis patients. The aim of this study is to investigate the effectiveness of virtual reality applications on balance, quality of life, and fall risk in postmenopausal osteoporosis patients and to compare them with a control group.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women aged 50-75 years
* Individuals diagnosed with osteoporosis based on Dual-Energy X-ray Absorptiometry (DEXA) measurement (T-score ≤ -2.5)
* Having been in menopause for at least 1 year
* Being able to walk independently (without the use of assistive devices)
* Volunteering to participate in the study and having provided informed consent
* Having adequate cognitive function (e.g., Mini Mental Test ≥ 24)

Exclusion Criteria:

* Secondary osteoporosis diagnosis (e.g. endocrine, metabolic or drug-induced causes)
* History of lower limb fracture or surgical intervention within the last 6 months
* Individuals with severe cardiovascular, neurological, or musculoskeletal disorders
* Individuals with vestibular or visual impairments that may affect balance
* Intolerance to virtual reality applications (e.g., dizziness, nausea, etc.)
* Individuals who have participated in a regular physiotherapy or exercise programme within the last 3 months

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-11-20 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Balance Level | 6 week
  Individual balance level assessments will be conducted using the Biodex balance device, which is reported to be valid and reliable for balance measurements, on both static and dynamic surfaces. The BDS consists of a mobile balance platform that provides a 360° range of motion and up to 20° surface inclination. The platform moves around the anteroposterior and mediolateral axes. The device measures the deviation of the centre of pressure in static conditions and calculates the degree of axis inclination in dynamic conditions. The difficulty level of the test is adjusted by changing the range of motion of the mobile platform and the surface inclination of the platform. Minimum stability on the platform can be set to 0 and maximum stability to 12. The test evaluates the patient's ability to maintain their centre of balance. The Biodex Balance System measures how far the patient's position deviates from the centre and reports the average deviation as a stability index. If the patient is
Cognitive State | 6 week
  The mini mental test, consisting of a total of 11 questions under five main headings: orientation, memory, attention and calculation, recall, and language, will be used to compare patients' cognitive status. This test is scored between 0 and 30. The assessment indicates that a score of 24-30 indicates normal cognitive function, 18-23 indicates mild cognitive impairment, and 18 points and below indicates that cognitive function is seriously impaired. A score of 24-30 indicates normal cognitive function, 18-23 indicates mild cognitive impairment, and 18 or below indicates that cognitive function is seriously impaired.
Risk of Falling | 6 week
  Individuals' risk of falling will be assessed using the BioDex balance device. The test measures the patient's postural sway velocity to predict the risk of falling. Speed is the individual's sway speed while maintaining balance. High scores suggest further evaluation for lower extremity strength, proprioception, and vestibular or visual deficits. In the fall risk test, individuals will stand upright with arms free on the BDS for 45 seconds with eyes open, then rest for 30 seconds. They will then wait for another 45 seconds with their eyes closed in the same upright standing position with arms free. The fall risk assessment results will be recorded as 'eyes open stance, eyes closed stance, and composite score'.

SECONDARY OUTCOMES:
Quality of life in patients | 6 week
  The QUALEFFO-41 quality of life questionnaire, which assesses osteoporosis-related quality of life and has been validated and proven reliable in Turkish; A; pain (5 questions), B; physical function/daily living activities (4 questions), C; physical function/household chores (5 questions), D; physical function/mobility (8 questions), E; social activities (7 questions), F; general health perception (3 questions), G; mental function (9 questions). Responses to the questions in the QUALEFFO-41 scale will be scored on a scale from 1 (healthy) to 5 (unhealthy).

CONTACTS AND LOCATIONS:
Overall Officials: İrem CANLI, Study Director — Kirsehir Ahi Evran Universitesi
Locations (1):
- Kırşehir Ahi Evran University, Merkez, Kirşehi̇r, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No